CLINICAL TRIAL: NCT05373316
Title: Addition of a Focal Boost in External Beam Radiotherapy for Locally Advanced Prostate Cancer by Online Adaptive MR-guided Radiotherapy
Acronym: AFFIRM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL79869.091.22
Record Dates: First submitted 2022-05-05; First posted 2022-05-13 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer; Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided hypofractionated focal boost radiotherapy (Experimental): External beam MR-guided (MR-linac) radiotherapy to the prostate and seminal vesicles of 5x7Gy (once weekly) with an isotoxic integrated focal boost up to 50Gy to the intraprostatic tumor as visible on multiparametric MR
  Interventions: Radiation: Ultrahypofractionated MR-guided radiotherapy boost

INTERVENTIONS:
Radiation: Ultrahypofractionated MR-guided radiotherapy boost — External beam MR-guided (MR-linac) radiotherapy to the prostate and seminal vesicles of 5x7Gy (once weekly) with an isotoxic integrated focal boost up to 50Gy to the intraprostatic tumor as visible on multiparametric MRI.

SUMMARY:
The AFFIRM trial tests the safety and clinical feasibility of MR-guided hypofractionated focal boost radiotherapy for patients with locally advanced prostate cancer. External beam radiotherapy combined with androgen deprivation therapy is considered as the treatment of choice for patients with locally advanced non-metastatic prostate cancer with seminal vesicle invasion.The long-term results of the multicentre phase III study (FLAME trial) showed that addition of an isotoxic focal boost to the intraprostatic lesion improves biochemical disease free survival in intermediate to high-risk patients without impacting toxicity and quality of life.

This focal boost strategy is now proven for a conventional fractionation scheme (35 fractions). The current trend in radiotherapy for prostate cancer is (extreme) hypofractionation, reducing the number of fractions. For locally advanced prostate cancer, however, the data on extreme hypofractionation are scarce.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or older with histologically proven prostate carcinoma
* Imaging stage T3b (as defined on mpMRI) N0M0
* Intraprostatic lesion visible on MRI
* Capable of giving informed consent

Exclusion Criteria:

* History of radiotherapy to the pelvis or transurethral resection of the prostate (TURP)
* Contraindications for MRI according to the guidelines of the local department of Radiology, inability to lay on a treatment table for 45-60 minutes or severe claustrophobia
* Absence of pre-treatment PSMA PET CT
* WHO performance score > 2
* International Prostate Symptom Score ≥ 15
* PSA > 30
* Prostate volume >100c

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Acute gastrointestinal and genitourinary toxicity | 90 days after start of treatment
  Acute gastrointestinal (GI) and genitourinary (GU) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Acute toxicity is defined as toxicity occurring within 90 days after the first radiation treatment (e.g. 60 days after completion of the radiation treatment).

SECONDARY OUTCOMES:
Late GI and GU toxicity (CTCAE v5.0) | from 90 days after start of treatment up to 5 years
  assessed between 90 days and up to 5 years after the first radiation treatment
Quality of life | from baseline up to 5 years after completion of treatment
  using the EORTC QLQ-C30 questionnaires
Quality of life | from baseline up to 5 years after completion of treatment
  using the EORTC QLQ-PR25 questionnaires
Biochemical disease free survival | up to 5 years after completion of treatment
  measuring the PSA concentration using the Phoenix definition for biochemical recurrence
Overall survival | up to 5 years after completion of treatment
Prostate cancer specific survival | up to 5 years after completion of treatment
Distant metastasis free survival | up to 5 years after completion of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Netherlands Cancer Institute, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Undecided